CLINICAL TRIAL: NCT06555263
Title: A Phase 2, Open-label Study Evaluating STRO-002, an Anti-folate Receptor Alpha (FOLR1) Antibody-Drug Conjugate, in Subjects With Previously Treated Advanced or Metastatic Non-small Cell Lung Cancer Expressing FOLR1
Brief Title: Study to Investigate Luveltamab Tazevibulin in Adults With Advanced or Metastatic Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated Early
Sponsor: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REFRaME-L1
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Lung Cancer, Nonsmall Cell; Lung Cancer Non-Small Cell Stage IIIB; Lung Cancer Non-small Cell Stage IV; Lung Cancer, Non-small Cell
Keywords: FOLR1; folate receptor alpha; FolRα; FRα; antibody drug conjugate; ADC; Luveltamab tazevibulin; STRO-002; Luvelta
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Luveltamab tazevibulin (Experimental): 4.3 mg/kg q3w
  Eligible subjects with stable disease (SD) may escalate to 5.2 mg/kg q3w after Cycle 4, with Sponsor approval.
  Interventions: Drug: Luveltamab tazevibulin

INTERVENTIONS:
Drug: Luveltamab tazevibulin — Luveltamab tazevibulin is an antibody-drug conjugate (ADC) targeting folate receptor α (FRα or FOLR1). It consists of an IgG1 antibody (SP8166) conjugated to cathepsin cleavable 3-aminophenyl hemiasterlin payload, yielding a homogenous ADC with a drug antibody ratio of four. The active warhead (SC209) inhibits tubulin polymerization leading to mitotic arrest and cell death.
  Other Names: STRO-002; luvelta

SUMMARY:
A Phase 2 study evaluating STRO-002 in subjects with previously treated advanced or metastatic non-small cell lung cancer expressing FOLR1

DETAILED DESCRIPTION:
This is a multicenter, open-label study. The study is designed to assess the preliminary efficacy and safety of luveltamab tazevibulin, an anti-FOLR1 antibody drug conjugate (ADC) in previously treated subjects with advanced or metastatic NSCLC that expresses FOLR1.

Subjects will receive luveltamab tazevibulin administered intravenously every 3 weeks until disease progression, intolerable toxicity, elective withdrawal from the study, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-squamous/adenocarcinoma or adenosquamous NSCLC that is either unresectable Stage IIIb/c disease not amenable for definitive chemoradiation, or Stage IV.
* Age ≥ 18 years
* ECOG performance status 0 to 1.
* Received at least 2 but no more than 4 prior lines of systemic therapy for advanced NSCLC
* Disease progression during or following the most recent systemic anti-cancer therapy.
* Positive FOLR1 expression per central testing
* At least 1 measurable target lesion per RECIST 1.1
* Adequate organ function

Exclusion Criteria:

* Prior treatment with a FOLR1- targeting ADCs or with ADCs that contain a tubulin inhibitor
* Untreated central nervous system metastases
* Ongoing immunosuppressive therapy, except for treated brain metastases, per criterion above.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or to antibody-related fusion protein treatment
* Pre-existing clinically significant ocular disorders, severe chronic obstructive pulmonary disease or asthma, clinically significant cardiac or cerebrovascular disease, or other significant concurrent, uncontrolled medical condition
* Previous solid organ transplantation
* Concurrent participation in another therapeutic treatment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  Best response of complete response (CR) or partial response (PR) per RECIST 1.1

SECONDARY OUTCOMES:
Duration of Response (DOR) per Investigator's assessment. | up to 24 months
  Confirmed CR or PR from the first documented response to the date of documented disease progression or death.
Progression Free Survival (PFS) by RECIST v1.1 per Investigator's assessment. | up to 24 months
  Time between the date of first dose and the first date of documented progression or death
Incidence and severity of adverse events and clinical laboratory abnormalities | up to 24 months
  Incidence and severity of adverse events (AEs) and clinical laboratory abnormalities.
ADC concentration | up to 24 months
  To evaluate the PK of luveltamab tazevibulin
Total antibody concentration | up to 24 months
  To evaluate the PK of luveltamab tazevibulin
Cytotoxic warhead concentration | up to 24 months
  To evaluate the PK of luveltamab tazevibulin

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UC San Diego Health - Moores Cancer Center, La Jolla, California
  - Georgetown University Medical Center - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute (FCS), Lake Mary, Florida
  - Tampa General Hospital - Cancer Center of South Florida, Tampa, Florida
  - HealthPartners Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Mary Crowley Cancer Research, Dallas, Texas